CLINICAL TRIAL: NCT01171976
Title: A 2 Year Randomized, Single-masked, Multicenter, Controlled Phase IIIb Trial Assessing the Efficacy and Safety of 0.5 mg Ranibizumab in Two "Treat and Extend" Treatment Algorithms vs. 0.5 mg Ranibizumab As Needed in Patients With Macular Edema and Visual Impairment Secondary to Diabetes Mellitus
Brief Title: Efficacy and Safety of Ranibizumab in Two "Treat and Extend" Treatment Algorithms Versus Ranibizumab As Needed in Patients With Macular Edema and Visual Impairment Secondary to Diabetes Mellitus
Acronym: RETAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRFB002D2304; 2010-019795-74 (EudraCT Number)
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Diabetic macula edema; RETAIN; ranibizumab
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- TE Ranibizumab 0.5 mg and Laser (Experimental): On Day 1, all patients received an intravitreal injection with 0.5 mg ranibizumab and subsequently entered Phase A which comprised of monthly injections. Laser therapy was applied at Day 1. It could then be re-administered according to ETDRS criteria at any visit with 0.5 mg ranibizumab treatment if deemed necessary by the Treating Investigator with a minimal treatment interval between laser treatments of 3 months. Laser therapy was administered ≥ 30 minutes prior to the ranibizumab injection.
  Interventions: Drug: Ranibizumab
- TE Ranibizumab 0.5 mg alone (Experimental): Patients received ranibizumab intravitreal injection therapy only.
  Interventions: Drug: Ranibizumab
- PRN Ranibizumab 0.5 mg (Active Comparator): Patients received ranibizumab intravitreal injection therapy as needed according to signs and symptoms of disease.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab (Lucentis®) was supplied in vials containing a dose of 0.5 mg/0.05 mL in an aqueous solution (pH 5.5) with histidine, trehalose, and polysorbate 20.

SUMMARY:
The purpose of this study is to demonstrate that two investigational treatment regimens have the potential to result in a superior visual acuity improvement as compared to a ranibizumab pro re nata (PRN=as needed) treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

Patient

* Patients with Type 1 or Type 2 diabetes mellitus (according to American Diabetes Association or World Health Organization [WHO] guidelines) with glycosylated hemoglobin (HbA1c) ≤ 12.0% at screening (Visit 1). Patients should be on diet, exercise, and/or pharmacological treatment for diabetes. Treatment for diabetes must have been stable for at least 3 month.

Ocular

* Patients with visual impairment due to DME in at least one eye who are eligible for laser treatment in the opinion of the investigator. If both eyes are eligible, the one with the worse visual acuity, as assessed at Visit 1, will be selected by the investigator as the study eye.
* BCVA ≥ 39 and ≤78 letters in the study eye and, inclusively, using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/160) at screening.
* Concomitant conditions in the study eye are only permitted if, in the opinion of the investigator, they do not prevent improvement of visual acuity on study treatment.

Exclusion Criteria:

Patient Compliance/ Administrative

* Pregnant or nursing (lactating) women.

Ocular medical history

* Active intraocular inflammation (grade trace or above) in either eye at enrollment.
* Any active infection (e.g. conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) in either eye at the time of enrollment.
* History of uveitis in either eye at any time.
* Structural damage within 0.5 disc diameter of the center of the macular in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema.
* Uncontrolled glaucoma in either eye at screening.

Prior Ocular treatments

* Panretinal laser photocoagulation in the study eye within 6 months prior to randomization.
* Focal/grid laser photocoagulation in the study eye within 3 months prior to randomization.
* Treatment with anti-angiogenic drugs in either eye.

Systemic conditions or treatments

* History of stroke within 6 months prior to enrollment.
* Renal failure requiring dialysis.
* Untreated diabetes mellitus.
* Blood pressure systolic > 160 mmHg or diastolic > 100 mmHg.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (61):
- Belgium (3):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
- Czechia (5):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
- France (8):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
- Greece (3):
  - Novartis Investigative Site, Heraklion Crete, Crete
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Győr
- Ireland (4):
  - Novartis Investigative Site, Dublin, Ireland
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Kilkenny
  - Novartis Investigative Site, Limerick
- Italy (3):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Netherlands (4):
  - Novartis Investigative Site, Leiden 2333 ZA, Netherlands
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
- Poland (4):
  - Novartis Investigative Site, Bielsko-Biala
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (3):
  - Novartis Investigative Site, Porto, Portugal
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
- Spain (8):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Zurich, Switzerland
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Binningen
- United Kingdom (10):
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, Aberdeen
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Sunderland
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] Prunte C, Fajnkuchen F, Mahmood S, Ricci F, Hatz K, Studnicka J, Bezlyak V, Parikh S, Stubbings WJ, Wenzel A, Figueira J; RETAIN Study Group. Ranibizumab 0.5 mg treat-and-extend regimen for diabetic macular oedema: the RETAIN study. Br J Ophthalmol. 2016 Jun;100(6):787-95. doi: 10.1136/bjophthalmol-2015-307249. Epub 2015 Oct 9. PMID 26453639

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 373 patients with macular edema and visual impairment secondary to DME were enrolled. A total of 372 patients were randomized. One patient was excluded from all analyses due to administrative problems
Pre-assignment Details: Antimicrobial eye drops were dispensed at each study visit (PRN ranibizumab) or at visits with scheduled injections (TE ranibizumab + laser or TE ranibizumab alone).
Groups:
- TE Ranibizumad 0.5 mg and Laser: Patients received an injection ranibizumab and laser therapy.
- TE Ranibizumab 0.5 mg Alone: Patients received an intravitreal injection ranibizumab
- PRN Ranibizumab 0.5 mg: Participants received ranibizumab intravitreal injection therapy as needed according to signs and symptoms of disease.
Period: Overall Study
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Started | 121 | 128 | 123
Safety Set | 126 (Include 4 from PRN and 3 from TE alone who got laser treatment, exclude 2 with no laser treatment.) | 126 (Exclude 1 who did not get drug and 3 got laser treatment, include 2 from 1st arm with no laser) | 118 (Exclude 1 who did not get drug and 4 got laser treatment)
Completed | 107 | 117 | 108
Not Completed | 14 | 11 | 15
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Death | 2 | 4 | 1
Not completed — Lost to Follow-up | 4 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 5 | 6
Not completed — Abnormal test result | 1 | 0 | 0
Not completed — Adverse Event | 6 | 2 | 5

BASELINE CHARACTERISTICS:
Population: The Randomized Set comprised all randomized patients, ie those given a randomization number.
Groups:
- Total: Total of all reporting groups
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg | Total
Number analyzed (Participants) | 121 | 128 | 123 | 372
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (9.07) | 63.0 (9.83) | 64.5 (9.66) | 63.7 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 51 | 46 | 140
  Male | 78 | 77 | 77 | 232

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity of the Study Eye: Average Change From Baseline to Month 1 Through Month 12
Description: Visual acuity was assessed at every study visit for the study eye using best correction determined from protocol refraction. The BCVA measurements were taken in a sitting position using ETDRS-like VA testing charts at a starting distance of 4 meters.
Time Frame: Baseline to Month 12
Population: Analyzed set included all randomized patients who received at least one application of study treatment and had at least one post baseline efficacy assessment. If missing values occurred without a subsequent observed value, the last observed value was carried forward to subsequent scheduled visits by means of a last observation carried forward.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Letters
  Baseline | 62.3 (11.50) | 64.1 (10.52) | 65.1 (10.08)
  Average Month 1 to Month 12 | 68.25 (11.057) | 70.28 (10.284) | 71.32 (9.984)
  Average Change from Baseline | 5.91 (5.532) | 6.14 (5.717) | 6.20 (6.005)

2. Secondary Outcome: Visual Acuity of the Study Eye: Average Change From Baseline to Month 1 Through Month 24
Description: as for outcome 1
Time Frame: Baseline to Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Letters
  Baseline | 62.3 (11.50) | 64.1 (10.52) | 65.1 (10.08)
  Average Month 1 to Month 24 | 69.12 (11.261) | 70.72 (10.924) | 72.09 (10.141)
  Average Change from Baseline | 6.78 (5.986) | 6.58 (7.070) | 6.97 (6.430)

3. Secondary Outcome: Visual Acuity of the Study Eye: Change From Baseline at Month 12
Description: as for outcome 1
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Letters
  Baseline | 62.3 (11.50) | 65.1 (10.52) | 65.1 (10.08)
  Month 12 | 69.13 (11.945) | 70.93 (11.742) | 72.56 (11.592)
  Change from Baseline | 6.79 (6.999) | 6.80 (8.726) | 7.44 (8.457)

4. Secondary Outcome: Visual Acuity of the Study Eye: Change From Baseline at Month 24
Description: as for outcome 1
Time Frame: Baseline and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Letters
  Baseline | 62.3 (11.50) | 64.1 (10.52) | 65.1 (10.08)
  Month 24 | 70.64 (12.315) | 70.62 (13.481) | 73.18 (11.872)
  Change from Baseline | 8.30 (8.129) | 6.49 (10.854) | 8.06 (8.462)

5. Secondary Outcome: Visual Acuity of the Study Eye: Categorized Change From Baseline at Month 12
Description: as for outcome 1
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Percentage of patients
  Gain of >= 1 letter | 82.9 | 84.8 | 83.8
  Gain of >= 5 letters | 59.0 | 60.8 | 70.1
  Gain of >= 10 letters | 32.5 | 42.4 | 39.3
  Gain of >= 15 letters | 19.7 | 30.4 | 26.5
  Loss of >= 5 letters | 3.4 | 4.0 | 3.4
  Loss of >= 10 letters | 0.0 | 2.4 | 0.9
  Loss of >= 15 letters | 0.0 | 1.6 | 0.9

6. Secondary Outcome: Visual Acuity of the Study Eye: Categorized Change From Baseline at Month 24
Description: as for outcome 1
Time Frame: Baseline, 24 month
Population: as for outcome 1
Measure: Number; unit: Percentage of pateints
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Percentage of pateints
  Gain of >= 1 letter | 87.2 | 84.0 | 90.6
  Gain of >= 5 letters | 69.2 | 62.4 | 76.1
  Gain of >= 10 letters | 43.6 | 40.8 | 45.3
  Gain of >= 15 letters | 25.6 | 28.0 | 30.8
  Loss of >= 5 letters | 4.3 | 8.0 | 5.1
  Loss of >= 10 letters | 2.6 | 7.2 | 3.4
  Loss of >= 15 letters | 0.9 | 4.0 | 2.6

7. Secondary Outcome: Central Subfield Thickness of the Study Eye: Percent Change From Baseline at Month 12
Description: High Resolution OCT was performed at every study visit by Spectral Domain OCT (if not available Time Domain OCT was acceptable) and the images were transferred to a digital video disc. These assessments were performed by trained and adequately qualified experts at the sites and prior to any study drug administration. CSFT is the average retinal thickness of the circular area with 1 mm diameter around the foveal center.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Percent Change | -27.09 (22.992) | -24.35 (22.027) | -23.16 (22.362)

8. Secondary Outcome: Central Subfield Thickness of the Study Eye: Percent Change From Baseline at Month 24
Description: as for outcome 7
Time Frame: Baseline and 24 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Percent Change | -32.03 (25.628) | -24.98 (26.414) | -24.97 (26.678)

9. Secondary Outcome: Visual Functioning Questionnaire (VFQ-25) Change From Baseline in Total Score at Month 12 and Month 24
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) was used to measure the influence of visual disability and symptoms on general health. The 12 subscales in the VFQ-25 are general health, general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision, and peripheral vision. For each, the patient was asked to rate their condition on a scale of 1-5 or 1-6, where a low number reflects a better outcome. Each response was recoded per the scoring rules outlined in the National Eye Institute (NEI) VFQ-25 Scoring Algorithm. Under this scoring algorithm , the recoded values range between 0 and 100 and a high score means a better functioning
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Score on a scale
  Baseline (n=116,122,114) | 75.32 (17.317) | 75.47 (17.105) | 77.07 (18.581)
  Change from baseline at Month 12 (n=116,122,114) | 4.60 (10.905) | 3.95 (10.941) | 5.41 (12.063)
  Change from baseline at month 24 (n=116,122,114) | 4.06 (11.859) | 2.31 (13.270) | 5.96 (12.389)

10. Secondary Outcome: EuroQoL (EQ-5D) Thermometer Score: Change From Baseline at Month 12 and Month 24
Description: The Euro Quality of Life Questionnaire (EQ-5D) is an indirect utility questionnaire. It is a standardized instrument was utilized to measure health outcomes related to 5 dimensions, namely: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The possible range for each dimension was 1 to 3, where 1= "no problems", 2="some problems" and 3="extreme problems" . A composite health index was then defined by combining the levels for each dimension. Overall, 243 health states are possible. For each health state, the EuroQol group has assigned a utility value typically between 0 and 1 with lower scores representing a higher level of dysfunction
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TE Ranibizumad 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Number analyzed (Participants) | 117 | 125 | 117
Score on a scale
  Baseline | 71.4 (17.36) [-2.18 to 2.69] | 70.7 (16.10) [-1.83 to 2.85] | 72.2 (13.24) [0.25 to 5.10]
  Change from Baseline at Month 12 (n=115,123,113) | 0.47 (16.487) [-1.11 to 4.00] | 0.91 (13.422) [-2.56 to 2.35] | 2.52 (14.431) [-0.11 to 4.97]
  Change from Baseline at Month 24 (n=115,123,113) | 1.35 (17.464) | 0.11 (14.755) | 1.98 (14.812)

ADVERSE EVENTS:
Description: The Safety Set consisted of all patients who received at least one administration of study treatment in the study eye and had at least one post-baseline safety assessment.
Groups:
- TE Ranibizumab 0.5 mg and Laser: Patients received an injection ranibizumab and laser therapy.
Arm/Group | TE Ranibizumab 0.5 mg and Laser | TE Ranibizumab 0.5 mg Alone | PRN Ranibizumab 0.5 mg
Serious Adverse Events (participants affected / at risk) | 34/126 | 29/126 | 26/118
Other Adverse Events (participants affected / at risk) | 98/126 | 101/126 | 78/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TE Ranibizumab 0.5 mg and Laser (N=126) | TE Ranibizumab 0.5 mg Alone (N=126) | PRN Ranibizumab 0.5 mg (N=118)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 4 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 2 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1
Cataract (Fellow eye) (Eye disorders) | 0 | 0 | 1
Macular fibrosis (Treated non-study eye) (Eye disorders) | 1 | 0 | 1
Vitreous adhesions (Treated non-study eye) (Eye disorders) | 0 | 0 | 1
Vitreous haemorrhage (Study eye) (Eye disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0
Small intestine ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 0
Bacterascites (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1 | 0
Endophthalmitis (Study eye) (Infections and infestations) | 1 | 0 | 0
Endophthalmitis (Treated non-study eye) (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0
Renal abscess (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Periorbital haematoma (Study eye) (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 3
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 1
Diabetic macroangiopathy (Vascular disorders) | 0 | 1 | 0
Diabetic vascular disorder (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TE Ranibizumab 0.5 mg and Laser (N=126) | TE Ranibizumab 0.5 mg Alone (N=126) | PRN Ranibizumab 0.5 mg (N=118)
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 4
Blepharitis (Study eye) (Eye disorders) | 2 | 1 | 0
Blindness transient (Study eye) (Eye disorders) | 0 | 2 | 0
Cataract (Fellow eye) (Eye disorders) | 3 | 4 | 2
Cataract (Study eye) (Eye disorders) | 5 | 7 | 7
Cataract (Treated non-study eye) (Eye disorders) | 2 | 3 | 1
Cataract subcapsular (Study eye) (Eye disorders) | 1 | 2 | 0
Conjunctival haemorrhage (Study eye) (Eye disorders) | 5 | 11 | 6
Conjunctival haemorrhage (Treated non-study eye) (Eye disorders) | 2 | 2 | 1
Conjunctivitis (Study eye) (Eye disorders) | 6 | 2 | 0
Corneal disorder (Study eye) (Eye disorders) | 2 | 0 | 0
Diabetic retinal oedema (Fellow eye) (Eye disorders) | 1 | 2 | 3
Diabetic retinal oedema (Study eye) (Eye disorders) | 4 | 2 | 1
Diabetic retinal oedema (Treated non-study eye) (Eye disorders) | 1 | 0 | 3
Diabetic retinopathy (Fellow eye) (Eye disorders) | 2 | 1 | 3
Dry eye (Fellow eye) (Eye disorders) | 3 | 0 | 3
Dry eye (Study eye) (Eye disorders) | 6 | 3 | 4
Dry eye (Treated non-study eye) (Eye disorders) | 2 | 1 | 1
Eye haemorrhage (Treated non-study eye) (Eye disorders) | 0 | 2 | 0
Eye irritation (Study eye) (Eye disorders) | 2 | 4 | 2
Eye pain (Fellow eye) (Eye disorders) | 2 | 0 | 2
Eye pain (Study eye) (Eye disorders) | 8 | 7 | 3
Eye pain (Treated non-study eye) (Eye disorders) | 1 | 0 | 2
Eye pruritus (Fellow eye) (Eye disorders) | 1 | 0 | 3
Eye pruritus (Study eye) (Eye disorders) | 2 | 2 | 2
Eye pruritus (Treated non-study eye) (Eye disorders) | 0 | 2 | 0
Eyelid oedema (Fellow eye) (Eye disorders) | 0 | 2 | 0
Eyelid oedema (Study eye) (Eye disorders) | 0 | 2 | 2
Foreign body sensation in eyes (Study eye) (Eye disorders) | 0 | 2 | 1
Glaucoma (Study eye) (Eye disorders) | 3 | 1 | 1
Keratitis (Study eye) (Eye disorders) | 1 | 3 | 0
Lacrimation increased (Study eye) (Eye disorders) | 1 | 4 | 0
Macular fibrosis (Fellow eye) (Eye disorders) | 2 | 0 | 1
Macular fibrosis (Study eye) (Eye disorders) | 3 | 0 | 0
Macular fibrosis (Treated non-study eye) (Eye disorders) | 3 | 1 | 2
Macular oedema (Fellow eye) (Eye disorders) | 3 | 6 | 3
Macular oedema (Study eye) (Eye disorders) | 2 | 3 | 2
Macular oedema (Treated non-study eye) (Eye disorders) | 1 | 3 | 0
Ocular hyperaemia (Study eye) (Eye disorders) | 2 | 1 | 1
Ocular hypertension (Fellow eye) (Eye disorders) | 3 | 1 | 2
Ocular hypertension (Study eye) (Eye disorders) | 7 | 2 | 3
Posterior capsule opacification (Fellow eye) (Eye disorders) | 1 | 0 | 2
Punctate keratitis (Study eye) (Eye disorders) | 2 | 0 | 2
Retinal exudates (Fellow eye) (Eye disorders) | 1 | 0 | 2
Retinal exudates (Study eye) (Eye disorders) | 0 | 2 | 2
Retinal haemorrhage (Study eye) (Eye disorders) | 2 | 3 | 0
Retinal haemorrhage (Treated non-study eye) (Eye disorders) | 2 | 1 | 0
Retinal neovascularisation (Fellow eye) (Eye disorders) | 1 | 4 | 3
Retinal vascular disorder (Study eye) (Eye disorders) | 2 | 0 | 0
Retinal vascular disorder (Treated non-study eye) (Eye disorders) | 2 | 0 | 0
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 2 | 2
Visual impairment (Study eye) (Eye disorders) | 0 | 0 | 2
Vitreous floaters (Study eye) (Eye disorders) | 0 | 1 | 4
Vitreous haemorrhage (Fellow eye) (Eye disorders) | 2 | 4 | 1
Vitreous haemorrhage (Study eye) (Eye disorders) | 8 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 7
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 4 | 3
Fatigue (General disorders) | 0 | 0 | 2
General physical health deterioration (General disorders) | 2 | 1 | 1
Influenza like illness (General disorders) | 3 | 0 | 1
Malaise (General disorders) | 0 | 1 | 2
Oedema peripheral (General disorders) | 7 | 5 | 3
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 3
Hypersensitivity (Immune system disorders) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 11 | 1 | 5
Bronchitis viral (Infections and infestations) | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 5 | 1
Conjunctivitis viral (Study eye) (Infections and infestations) | 2 | 0 | 0
Cystitis (Infections and infestations) | 2 | 2 | 6
Ear infection (Infections and infestations) | 1 | 1 | 3
Gastroenteritis (Infections and infestations) | 2 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 3 | 1
Hordeolum (Study eye) (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 9 | 10 | 8
Laryngitis (Infections and infestations) | 0 | 1 | 2
Localised infection (Infections and infestations) | 2 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 3 | 3
Nasopharyngitis (Infections and infestations) | 11 | 10 | 8
Paronychia (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 3 | 1
Skin infection (Infections and infestations) | 0 | 3 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 2
Tooth infection (Infections and infestations) | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 4
Urinary tract infection (Infections and infestations) | 9 | 10 | 5
Viral infection (Infections and infestations) | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 3 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 4
Blood bilirubin increased (Investigations) | 0 | 2 | 1
Blood creatinine increased (Investigations) | 2 | 4 | 0
Blood glucose increased (Investigations) | 2 | 3 | 3
Blood lactate dehydrogenase increased (Investigations) | 1 | 4 | 3
Blood potassium increased (Investigations) | 3 | 4 | 2
Blood urea increased (Investigations) | 3 | 4 | 2
Blood uric acid increased (Investigations) | 3 | 2 | 1
Blood urine present (Investigations) | 2 | 3 | 4
Gamma-glutamyltransferase increased (Investigations) | 3 | 6 | 4
Glycosylated haemoglobin increased (Investigations) | 0 | 2 | 2
Haematocrit decreased (Investigations) | 1 | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 4 | 1
Intraocular pressure increased (Fellow eye) (Investigations) | 2 | 2 | 1
Intraocular pressure increased (Study eye) (Investigations) | 2 | 7 | 5
Platelet count decreased (Investigations) | 1 | 1 | 3
Protein total increased (Investigations) | 1 | 1 | 2
Red blood cell count decreased (Investigations) | 1 | 2 | 0
White blood cell count increased (Investigations) | 1 | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 3 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 4 | 4
Gout (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 3 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 4 | 1
Ketosis (Metabolism and nutrition disorders) | 0 | 1 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 10 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Diabetic neuropathy (Nervous system disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 2 | 2
Headache (Nervous system disorders) | 4 | 1 | 4
Hypoglycaemic coma (Nervous system disorders) | 2 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 2
Sciatica (Nervous system disorders) | 2 | 1 | 2
Syncope (Nervous system disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 2 | 3
Insomnia (Psychiatric disorders) | 4 | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 2 | 1
Renal impairment (Renal and urinary disorders) | 2 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 19 | 17 | 8
Hypotension (Vascular disorders) | 1 | 2 | 0
Venous insufficiency (Vascular disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of the pooled data (i.e. data from all sites) in the clinical trial or disclosure of trial results in their entirety.